CLINICAL TRIAL: NCT00450879
Title: Pilot Study of GW786034 (Pazopanib), a Vascular Endothelial Growth Factor Receptor Tyrosine Kinase Inhibitor, in Patients With Operable Breast Cancer
Brief Title: Pazopanib in Treating Patients With Newly Diagnosed or Locally and/or Regionally Recurrent Breast Cancer That Can Be Removed By Surgery
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00183; NCI-2009-00183 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000534258; 040607; 040607 (Other: Rutgers Cancer Institute of New Jersey); 7529 (Other: CTEP); U01CA132194 (NIH); P30CA072720 (NIH)
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2013-06

CONDITIONS: Male Breast Carcinoma; Recurrent Breast Carcinoma; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer; Stage IIIA Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — pazopanib

ARMS (1):
- Treatment (pazopanib hydrochloride) (Experimental): Patients receive pazopanib hydrochloride PO QD for 12-20 days in the absence of disease progression or unacceptable toxicity. Patients then undergo surgical resection of tumor between days 13 and 21 (24 hours after completion of pazopanib hydrochloride).
  Interventions: Drug: Pazopanib Hydrochloride; Procedure: Dynamic Contrast-Enhanced Magnetic Resonance Imaging; Other: Pharmacological Study; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Pazopanib Hydrochloride — Given PO
  Other Names: GW786034B; Votrient
Procedure: Dynamic Contrast-Enhanced Magnetic Resonance Imaging — Correlative studies
  Other Names: DCE MRI; DCE-MRI
Other: Pharmacological Study — Correlative studies
  Other Names: pharmacological studies
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This pilot clinical trial studies how well pazopanib hydrochloride works in treating patients with breast cancer that is newly diagnosed or has come back at or near the same place as the original tumor and can be removed by surgery. Pazopanib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by preventing the growth of new blood vessels necessary for tumor growth. Giving pazopanib hydrochloride before surgery may make the tumor smaller and reduce the amount of tissue that needs to be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the biologic effect, measured by a decrease in phosphorylation of vascular endothelial growth factor receptor 2 (VEGFR-2) and/or decrease in microvessel density, in breast tumor biopsies after treatment with daily oral GW786034 (pazopanib hydrochloride) for at least 12 consecutive days in early stage, operable breast cancer or local and/or regional recurrence that is amenable to surgery.

II. To determine the mechanism of antitumor effect, measured by a reduction in tumor cell proliferation (Ki67) or an increase in apoptosis in breast tumor biopsies after treatment with GW786034.

SECONDARY OBJECTIVES:

I. To determine the change in levels of tissue vascular endothelial growth factor (VEGF) in breast tumor biopsies after treatment with GW786034.

II. To evaluate the change in phosphorylation of epidermal growth factor receptor (EGFR), mitogen-activated protein kinase (MAPK), and protein kinase B (AKT) in breast tumor biopsies after treatment with GW786034.

III. To identify gene expression patterns in breast tumor biopsies before and after treatment with GW786034.

IV. To evaluate the change in VEGF (in the plasma) and VEGFR-2 (in the serum) as circulating biomarkers after treatment with GW786034.

V. To evaluate the change in circulating tumor cells in peripheral blood after treatment with GW786034.

VI. To determine whether the steady-state plasma concentration of GW786034 correlates with inhibition of phosphorylated (phospho)-VEGFR-2 and other endpoints in breast tumor biopsies.

VII. To evaluate the change in vascular permeability by dynamic contrast enhanced (DCE)-magnetic resonance imaging (MRI) of the breast after treatment with GW786034.

VIII. To compare the images obtained with bilateral DCE-MRI of the breast before, during, and after treatment with GW786034.

OUTLINE:

Patients receive pazopanib hydrochloride orally (PO) once daily (QD) for 12-20 days in the absence of disease progression or unacceptable toxicity. Patients then undergo surgical resection of tumor between days 13 and 21 (24 hours after completion of pazopanib hydrochloride).

After completion of study treatment, patients are followed up within 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of invasive adenocarcinoma of the breast by core needle biopsy or limited incisional biopsy
* Tumor size >= 1.0 cm as assessed by physical exam or radiographic exam
* Patients with histologically verified local and/or regional recurrence of invasive breast cancer that is amenable to surgery and meet all eligibility criteria may participate
* No prior chemotherapy or hormonal therapy for this primary breast cancer
* Patients who can undergo surgical treatment with either lumpectomy or mastectomy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* White blood cells (WBC) >= 3,000/uL
* Platelets >= 100,000/uL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x institutional upper limit of normal (ULN)
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Prothrombin time (PT)/international normalized ratio (INR)/partial thromboplastin time (PTT) =< 1.2 x institutional ULN
* Urine protein:creatinine ratio (UPC) of less than or equal to 1 as assessed in a random or spot urine sample
* Patients must have blood pressure (BP) no greater than 140 mmHg (systolic) and 90 mmHg (diastolic) for eligibility; initiation or adjustment of BP medication is permitted prior to study entry provided that the average of three BP readings at a visit prior to enrollment is less than 140/90 mmHg
* Eligibility of patients receiving any medications or substances known to affect or with the potential to affect the activity or pharmacokinetics of GW786034 (pazopanib) will be determined following review of their case by the Principal Investigator
* Women of child-bearing potential and men must agree to use adequate contraception (barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should (barrier method of birth control; abstinence)
* Any concomitant medications that are associated with a risk of QTc prolongation and/or Torsades de Pointes should be discontinued or replaced with drugs that do not carry these risks, if possible; patients who must take medications with a risk or possible risk of Torsades de Pointes should be watched carefully for symptoms of QTc prolongation, such as syncope

Exclusion Criteria:

* Patients with locally advanced breast cancer who are not candidates for surgical resection at time of initial evaluation, this may include patients with locally advanced disease such as:

  * Tumor of any size with direct extension to chest wall or skin (T4a-c)
  * Inflammatory breast cancer (T4d)
* Patients with evidence of metastatic disease
* Patients may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to GW786034 (pazopanib) or other agents used in the study are excluded
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with a baseline QTc >= 480 msecs or other significant electrocardiogram (ECG) abnormalities are ineligible
* Patients with poorly controlled hypertension (systolic blood pressure of 140 mmHg or higher, or diastolic blood pressure of 90 mmHg or higher) are ineligible
* Certain medications that act through the cytochrome p 450 (CYP450) system are specifically prohibited in patients receiving GW786034 (pazopanib); certain other agents should be used with caution
* Patients with any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for intravenous [IV] alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease) that impairs their ability to swallow and retain GW786034 (pazopanib) tablets are excluded
* Patients with any of the following conditions are excluded:

  * Serious or non-healing wound, ulcer, or bone fracture
  * History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days of treatment
  * Any history of cerebrovascular accident (CVA) within the last 6 months
  * Current use of therapeutic warfarin; Note: Low molecular weight heparin and prophylactic low-dose warfarin are permitted; PT/PTT must meet the inclusion criteria * History of myocardial infarction, cardiac arrhythmia, admission for unstable angina, cardiac angioplasty or stenting within the last 12 weeks
  * History of venous thrombosis in last 12 weeks
  * Class III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system; a patient who has a history of class II heart failure and is asymptomatic on treatment may be considered eligible
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situation that would limit compliance with study requirements
* Pregnant women are excluded from this study; procedures affecting absorption, or active peptic ulcer disease) that impairs their ability to swallow and retain GW786034 (pazopanib) tablets are excluded
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Inability to understand or unwillingness to sign a written informed consent document

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-01; Primary Completion 2010-11 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Change in molecular parameters such as phosphorylated VEGFR-2, microvessel density, tumor proliferation (Ki67), and apoptosis | Baseline to up to 20 days
  The pre-post comparison of the biologic effects in the tumor can be done by a paired t-test as they are all continuous variables. If the differences are not normally distributed, transformations or non-parametric methods will be applied. Multiple comparisons will be adjusted for using Bonferroni method as the biologic effects are measured by four variables. The relationship among these four variables will be analyzed using factor analysis to see if they can be reduced to one or two representative indices.

SECONDARY OUTCOMES:
Change in plasma VEGF levels | Baseline to up to 20 days
  The pre-post difference of the tissue variables will be regressed on the plasma VEGF levels.
Change in serum VEGFR-2 levels | Baseline to up to 20 days
  The pre-post difference of the tissue variables will be regressed on the serum VEGFR-2 levels.
Change in circulating tumor cells | Baseline to up to 20 days
Stead-state plasma concentration of pazopanib hydrochloride | Baseline (pre-dose day 1), day 8, and 24-72 hours prior to surgery
  The pre-post difference of the tissue variables will be regressed on the plasma concentration of pazopanib hydrochloride.
Change in images obtained with bilateral DCE-MRI of the breast | Baseline to up to 20 days

CONTACTS AND LOCATIONS:
Overall Officials: Antoinette Tan, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States